CLINICAL TRIAL: NCT01152398
Title: A Phase I Safety and Immunogenicity Trial of MVA-BN®-HER2 Vaccine in HER-2-Positive Breast Cancer Patients Following Adjuvant Therapy
Brief Title: A Safety and Immunology Study of a Modified Vaccinia Vaccine for HER-2(+) Breast Cancer After Adjuvant Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNIT-BR-003; NCT01158469 (obsolete NCT alias)
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2011-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Vaccine; Metastatic; HER-2-positive; Phase I; HER-2 Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MVA-BN-HER2 (Experimental)
  Interventions: Biological: MVA-BN-HER2

INTERVENTIONS:
Biological: MVA-BN-HER2 — experimental vaccine, subcutaneous injection q4weeks x6

SUMMARY:
The current trial, BNIT-BR-003, will evaluate the safety and biological activity of a fixed dose of MVA-BN®-HER2 following adjuvant chemotherapy in patients with HER-2-positive breast cancer.

The intent of vaccination is to induce a combined antibody and T-cell anti-HER-2 immune response, which is intended to target HER-2-expressing tumor cells, and may induce tumor regression or slow progression of disease.

DETAILED DESCRIPTION:
MVA-BN®-HER2 is a candidate breast cancer immunotherapy product comprised of a highly attenuated non-replicating vaccinia virus, MVA-BN®, engineered to encode a modified form of the HER-2 protein.

MVA-BN® is a well-characterized, clonal strain of modified vaccinia virus Ankara (MVA) being developed as a smallpox vaccine, suitable for use in high-risk (e.g., immunocompromised) individuals. MVA-BN®-derived vectors encoding heterologous antigens are being developed for use as vaccines for infectious diseases such as HIV, and for the treatment of cancer. A large database exists from safety evaluations in animals and in humans for MVA-BN®, and MVA-BN®-derived vectors.

HER-2 is overexpressed in 20-30% of human breast cancers. It is an oncogene/growth factor receptor critical for the malignant phenotype of HER-2- expressing tumors. It is an immunogenic target, and immune responses to this protein have been shown to mediate potent anti-tumor activity in multiple animal models. Means to stimulate anti-HER-2 reactivity are now being studied clinically. Sponsor, collaborators, and others have used both Protein and DNA vaccine forms of HER-2, and a safety database is developed and no significant adverse events have resulted from HER-2 directed vaccination.

MVA-BN®-HER2 encodes a modified form of the HER-2 protein, hereinafter referred to as HER2. HER2 contains the extracellular domain of HER-2 but lacks the intracellular, cell signaling domain. In addition, HER2 includes two universal T-cell epitopes from tetanus toxin to facilitate the stimulation of an immune response to HER-2, a self-protein.

The current trial, BNIT-BR-003, will evaluate the safety and biological activity of a fixed dose of MVA-BN®-HER2 following adjuvant chemotherapy in patients with breast cancers which overexpress HER-2.

Patients will receive 6 subcutaneous vaccinations at 4-week intervals and will have blood drawn for immune function analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Women, ≥ 18 years of age
* Histologically documented, HER-2-positive breast cancer without metastatic disease. Hormone receptor (ER/PR) status may be either positive or negative. HER-2 (+) status may be determined by one of the following measurements:
* Immunohistochemistry 3+ or FISH/CISH+ (HER-2 gene signal to centromere 17 signal > 2). NOTE: HER-2 assessment may have been on initial diagnosis and need not be repeated.
* Patients should be assessed as having no evidence of disease (NED) at the end of adjuvant chemotherapy. In addition, these patients must have a clinical evaluation and lab work as standard of care disease assessment without evidence of recurrence within 28 days of the first planned dose of MVA-BN®-HER2.
* Completed adjuvant and/or neoadjuvant chemotherapy for breast cancer at least 3 months previously (measured from the date of the last dose of chemotherapy) and prior to the first planned dose of MVA-BN®-HER2).
* ECOG Performance Score of 0, 1.
* Predicted life expectancy ≥ 12 months
* Left ventricular ejection fraction (LVEF) by ECHO ≥ LLN as defined by institutional standards
* Women of childbearing potential must:

  * have a negative serum or urine pregnancy test, and
  * must agree to use a medically acceptable barrier and/or chemical method of contraception throughout the study treatment period and for 28 days after the last dose of MVA-BN®-HER2.
* No significant cardiac, bone marrow dysfunction, or coagulopathy (defined as no Grade 3 or greater AE according to NCI CTCAE v 3.0). No significant hepatic or renal dysfunction (defined as no Grade 2 or greater AE according to NCI CTCAE v 3.0. Patients with a known history of a CLINICALLY NON-SIGNIFICANT laboratory parameter may be eligible for inclusion provided an exemption is granted by the study Medical Monitor prior to enrollment.
* A negative virology screen for HIV, HBsAg, and HCV

Exclusion Criteria:

* Congestive heart failure (NYHA Class III or IV), unstable angina, or cardiovascular disease such as stroke or myocardial infarction (current or within the past 6 months)
* History of cardiac toxicity secondary to chemotherapy or Herceptin immunotherapy (LVEF decline of 15% or greater from baseline)
* History of prior malignancies other than breast cancer within the past 5 years, excluding basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Any breast cancer metastases beyond the lymph nodes
* Known allergy to eggs, egg products, or aminoglycoside antibiotics, e.g., gentamicin or tobramycin
* Chronic administration (defined as 6 or more consecutive days of use) of systemic corticosteroids within 14 days of the first planned dose of MVA-BN®-HER2. Limited use of inhaled steroids, nasal sprays, eye drops, and topical creams for small body areas is allowed.
* History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement hormones are not excluded.
* Prior solid organ or hematopoietic allogenic transplant(s)
* Prior use of hematopoietic growth factors (e.g., GM-CSF) within 14 days of the first planned dose of MVA-BN®-HER2
* Receipt of an investigational agent within 28 days of the first planned dose of MVA-BN®-HER2
* Prior "vaccine" therapy for breast cancer at any time
* Vaccination:

Live (attenuated) vaccine (e.g., FluMist®) Vaccination with a live vaccine within 28 days of the first planned dose of MVA-BN®-HER2, or plans to receive a live vaccine within 28 days after the last dose of MVA-BN®-HER2 is not allowed Killed (inactivated) vaccine (e.g.,PneumoVax®) Vaccination with a killed vaccine within 14 days of the first planned dose of MVA-BN®-HER2, or plans to receive a killed vaccine within 14 ' days after the last dose of MVA-BN®-HER2 is not allowed

* A maximum cumulative dose of prior doxorubicin > 360 mg/m2 or epirubicn > 720 mg/m2
* Radiation therapy within 14 days of the first planned dose of MVA-BN®-HER2 or plans for radiation therapy after enrollment. Prior to initiating palliative radiation during the treatment phase of the study, the Sponsor's medical monitor or designee must be contacted.
* Pregnant, lactating, or nursing
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial or the long-term follow-up study, or would interfere with the evaluation of the trial endpoints

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number and type of adverse events as a measure of safety and tolerability of multiple vaccinations | 18 months

SECONDARY OUTCOMES:
Type and duration of immune response measured over time to repeat vaccine administrations | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bandman, Study Director — Bavarian Nordic
Locations (1):
- Alta Bates Comprehensive Cancer Center, Berkeley, California, United States